CLINICAL TRIAL: NCT02831556
Title: A Pilot Study to Test Rapid Acquisition of Point of Care Ultrasound for Various Applications
Brief Title: Point of Care 3D Ultrasound for Various Applications: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00071789
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Appendicitis; Evidence of Cholecystectomy; Gallstones; Pregnancy, Ectopic; Aortic Aneurysm; Kidney Stones; Intrauterine Pregnancy; Diverticulitis; Abdominal Injuries; Tumors; Pancreatitis; Digestive System Diseases; Gastrointestinal Diseases; Intraabdominal Infections; Intestinal Diseases; Pregnancy; Vascular Disease; Uterine Fibroids; Ovarian Cysts; Uterine Abnominalies; Bladder Abnominalies; Testicular Abnominalies; Polyps
Keywords: Ultrasound; Abdomen; Pelvis; 3D
MeSH Terms: conditions — Appendicitis; Gallstones; Pregnancy, Ectopic; Aortic Aneurysm; Kidney Calculi; Diverticulitis; Abdominal Injuries; Neoplasms; Pancreatitis; Digestive System Diseases; Gastrointestinal Diseases; Intraabdominal Infections; Intestinal Diseases; Vascular Diseases; Leiomyoma; Ovarian Cysts; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Emergency Department Subjects: Subjects that present to the Emergency Department with complaints necessitating abdominal or pelvic imaging.
- Non-patient volunteers: Duke employees that will voluntarily have an abdominal or pelvic ultrasound for with the sole purpose being for the study.

SUMMARY:
Summary

1. Purpose and Objective: The purpose of this study is to test the feasibility of rapid acquisition of point of care 3D ultrasound in obtaining abdominal and/or pelvic images. The study will use a newly developed acquisition method and post-processing technique to create three dimensional image models of the abdomen and/or pelvis.
2. Study activities and population group. The study population will be a convenience sample of patients of any age presenting to the Emergency Department with complaints necessitating a clinical abdominal and/or pelvic imaging. The study intervention includes acquisition of research ultrasound images, which will not be used for clinical care, and comparison of these images with clinically obtained images. Other clinical data such as surgical and pathology reports will also be reviewed. 3.Data analysis and risk/safety issues. This is a pilot study intended to determine feasibility and to refine image reconstruction algorithms. Research images will be compared to clinical images. Comparison of research images with final diagnosis will also occur. The research intervention, an ultrasound exam, has no known safety risks. The only risk to subjects is loss of confidentiality.

This study is observational, not interventional, because the experimental ultrasound will be performed in all subjects and will not be used in the clinical care of patients (consequently, will not have the opportunity to affect clinical outcomes). Experimental images will be reviewed after completion of clinical care and will not be provided to the clinicians caring for the subjects. The investigators are not measuring the effect of the ultrasound examination on the subjects' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must present to the emergency department for evaluation of complaints suspected to be related to an abdominal or pelvic pathology. The clinical diagnostic plan before subject enrollment may include abdominal or pelvic ultrasound, CT scan and/or MRI.

OR

* Non-patient volunteer

Exclusion Criteria:

* Non-English speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age that present to the Emergency Department with chief complaints suspected to be related to an abdominal or pelvic pathology for which clinical imaging is ordered.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2016-07; Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Experimental ultrasound diagnosis agreement with final reference standard diagnosis | Comparison of experimental ultrasound diagnosis with final reference diagnosis will occur at approximately 4 weeks (average) after date of experimental ultrasound exam, to allow clinical follow-up to occur.

SECONDARY OUTCOMES:
Duration of experimental ultrasound exam | The duration of the experimental ultrasound exam in seconds will be digitally recorded at the time of its performance. We anticipate the ultrasound duration to be less than 600 seconds
Experimental ultrasound image quality. | 4 weeks (average). Images will be reviewed after the completion of each subject's acute care. Image review will usually occur within 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Broder, MD, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No